CLINICAL TRIAL: NCT00044668
Title: An Open-Label Study to Examine the Long-Term Effect on Glucose Control (HbA1c) and Safety of AC2993 Given Two Times a Day to Subjects With Type 2 Diabetes Treated With Metformin, a Sulfonylurea, or Metformin and Sulfonylurea Combination
Brief Title: Evaluation of the Effect on Glucose Control and Safety of AC2993 in Patients With Type 2 Diabetes Treated With Metformin, Sulfonylurea, or Metformin and Sulfonylurea Combination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2993-117
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: exenatide; exendin-4; diabetes; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AC2993 (Experimental): 5 μg AC2993, twice daily, for 4 weeks followed by 10 μg AC2993, twice daily, during a maintenance period
  Interventions: Drug: AC2993

INTERVENTIONS:
Drug: AC2993 — Subjects will receive 5 μg AC2993, subcutaneously injected twice daily, for 4 weeks followed by 10 μg AC2993, subcutaneously injected twice daily, during a maintenance period that is expected to continue for at least 11 months.
  Other Names: synthetic exendin-4

SUMMARY:
This multi-center, open-label study is designed to examine the effects on long-term glucose control and safety of AC2993 in patients with type 2 diabetes treated with metformin, sulfonylurea, or metformin and sulfonylurea combination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* Treated for at least 3 months prior to screening either with metformin, sulfonylurea, or metformin and sulfonylurea combination
* BMI 25-45 kg/m^2
* HbA1c between 7.5 % and 12.0 %, inclusive

Exclusion Criteria:

* Treated with other oral anti-diabetic agents other than metformin and sulfonylureas within 3 months of screening
* Patients previously treated with AC2993
* Patients presently treated with insulin

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2002-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Baseline to Week 24, Week 52, and to each intermediate visit | Baseline, and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
  Change in HbA1c from Baseline to Week 24, Week 52, and to each intermediate visit (Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52)
Change in concentrations of fasting plasma glucose and lipids from Baseline Visit 2 (Day 1) to Week 24, to Week 52, and to each intermediate visit | Baseline, and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
  Change in concentrations of fasting plasma glucose and lipids from Baseline Visit 2 (Day 1) to Visit 10 (Week 24), to Visit 14 (Week 52) and to each intermediate visit (Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (3):
- Hungary (3):
  - Diagnostic Units Hungary Kft., Budapest, Hungary
  - Peterfy Teaching Hospital, Budapest, Hungary
  - Uzsoki Street Municipal Hospital, Budapest, Hungary

REFERENCES:
- [Derived] Ivanyi T, Fovenyi J, Faludi P, Han J, Macconell L, Wille S, Kiljanski J. Long-term effects of adding exenatide to a regimen of metformin and/or sulfonylurea in type 2 diabetes: an uncontrolled, open-label trial in Hungary. Clin Ther. 2012 Jun;34(6):1301-13. doi: 10.1016/j.clinthera.2012.04.022. Epub 2012 May 16. PMID 22608106
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356